CLINICAL TRIAL: NCT01248520
Title: Text Messaging For Preventative Health During Pregnancy; Improving Influenza Vaccination Rates In Pregnancy: A Randomized Controlled Trial of Text Messaging to Increase Vaccine Uptake
Brief Title: Influenza and Text Messaging in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Richard Beigi, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO09100504
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Pregnancy
Keywords: Pregnancy; Influenza Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- General health information (Placebo Comparator): Pregnant women receiving text messages containing general health messages without including information regarding the importance of the influenza vaccination
  Interventions: Other: general health information
- Influenza and general health information (Active Comparator): Pregnant women receiving text messages with influenza facts and the importance of the influenza vaccination, as well as general health messages Intervention: Text messages with influenza facts
  Interventions: Other: influenza and general health information

INTERVENTIONS:
Other: influenza and general health information — Subjects assigned to the influenza information group will receive health text messages from the time they enroll until they deliver. These messages will contain general health information as well as information regarding influenza and the importance of vaccination during pregnancy.
  Arms: Influenza and general health information
Other: general health information — Subjects assigned to the influenza information group will receive health text messages from the time they enroll until they deliver.
  Arms: General health information

SUMMARY:
A randomized, controlled clinical trial to assess whether text messaging to an outpatient obstetric population can improve maternal influenza vaccine uptake.

DETAILED DESCRIPTION:
History and the 2009 H1N1 influenza pandemic suggest that both seasonal and pandemic influenza infections impart disproportionate morbidity and mortality among gravidas. The influenza vaccine represents a viable, preventive health intervention to mitigate disease burden for gravidas and their neonates. Despite the safety and efficacy of influenza vaccines, suboptimal maternal vaccination rates (13-24%) persist nationwide. Barriers to influenza vaccination during pregnancy include patient concerns about vaccine safety and unappreciated risk of influenza infection. Cellular phone text messaging has emerged as an innovative technology with advantages of ubiquity, rapid, confidential information transmission, and low cost. Text messaging may represent an effective way to educate pregnant women about their particular vulnerability to influenza infection and enhance influenza vaccine uptake. We propose a randomized, controlled clinical trial to assess whether text messaging to an outpatient obstetric population can improve maternal influenza vaccine uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women less than 28 weeks estimated gestation age
2. Between 14-50 years of age
3. Willing to provide informed consent and undergo necessary study procedures

Exclusion Criteria:

1. Unwillingness or inability to receive text messages
2. Receipt of the current season's influenza vaccine or plan to receive the influenza vaccine on the day of the enrollment visit
3. Reported history of adverse reaction precluding receipt of the vaccine
4. Unwillingness or inability to provide informed consent and comply with study criteria.

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To assess the ability of direct communication and education to patients using modern technology (cellular text messaging) to enhance vaccine uptake. | at participant post-partum visit
  To assess the ability of direct communication and education to patients using modern technology (cellular text messaging) to enhance vaccine uptake. We hypothesize that text messaging will improve the timing (earlier in flu season) and rate of receipt of influenza vaccination in pregnancy.

SECONDARY OUTCOMES:
To assess the ability of direct education via text messaging to enhance knowledge about influenza infection and vaccination in pregnancy. | at participant post-partum visit
  To assess the ability of direct education via text messaging to enhance knowledge about influenza infection and vaccination in pregnancy. We hypothesize that women receiving text messages will be more likely than controls to have accurate knowledge about pregnant women's increased susceptibility to influenza and about the vaccine's safety and efficacy in pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Moniz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moniz MH, Hasley S, Meyn LA, Beigi RH. Improving influenza vaccination rates in pregnancy through text messaging: a randomized controlled trial. Obstet Gynecol. 2013 Apr;121(4):734-740. doi: 10.1097/AOG.0b013e31828642b1. PMID 23635672